CLINICAL TRIAL: NCT04730167
Title: The Monaco Initiative for Concussion in Motorsport Pilots: Brain Exploration in Retired Motorsport Pilots
Brief Title: The Monaco Initiative for Concussion in Motorsport Pilots
Status: Completed | Type: Observational
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other); University of Cambridge (Other); Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Other Study IDs: MIMP
Record Dates: First submitted 2021-01-19; First posted 2021-01-29 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-05

CONDITIONS: Brain Injuries; Concussion, Brain; Sport Injury
Keywords: Motorsport Pilots; Concussions; Brain trauma; Traumatic brain injuries; MRI; positron emission tomography (PET) scan; Video-oculography; Oculomotor behaviors
MeSH Terms: conditions — Brain Injuries; Brain Concussion; Brain Injuries, Traumatic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retired Motorsport Pilots: Concussion assessment
  Interventions: Other: Neurological and neuropsychological assessments / MRI / PET scan / Video-oculography.

INTERVENTIONS:
Other: Neurological and neuropsychological assessments / MRI / PET scan / Video-oculography. — Essential data for this study are those collected during the concussion assessment, carried out as part of routine care at Princess Grace Hospital (medical background; history of sports practice and history of concussions; data extracted from clinical and neuropsychological evaluations, from imaging exams (MRI and PET-Scan) and from eye-tracking evaluation).

SUMMARY:
The study aims:

* to observe a population particularly exposed by the past to brain trauma and concussion: Motorsport Pilots who are retired from a professional practice of motor sport;
* to report results of their neuro-cognitive evaluations,
* to determine if specific profiles emerge.
* to evaluate potential consequences of these traumas' history at a cerebral, physical and psychological level.
* to evaluate the contribution of the various examinations performed as part of a concussion assessment in routine care (eye-tracking, brain imaging, Neuropsychological Assessment).

DETAILED DESCRIPTION:
The Memory Center of the Rainier III Center and The Department of Nuclear Medicine of the Princess Grace Hospital are particularly aware of evaluation, management and monitoring of patients who have suffered brain trauma, or concussions, and the study of possible long-term consequences.

They regularly receive patients, referred by neurologists or spontaneously coming for consultation, for whom the carrying out of a complete in-depth evaluation is recommended, because of their medical history and their personal history.

In partnership with the "Fédération Internationale de l'Automobile" (FIA) and the "Automobile Club of Monaco" (ACM), the Princess Grace Hospital team hopes ultimately to set up a screening campaign for traumatic brain injuries among a particularly exposed population: motorsports people.

In this context, inspired by the work carried out by the Cambridge University team (the Rescue Racer Study) and the FIA recommendations, the Sponsor wishes to carry out an observational study with retired motor sportspeople.

The objectives are to study a population particularly exposed by the past to brain trauma and concussion (who is retired from a professional practice of motor sport), to report results of their neuro-cognitive evaluations, and to determine if specific profiles emerge, to evaluate potential consequences of these traumas' history at a cerebral, physical and psychological level.

ELIGIBILITY:
* Men or women.
* Aged 18 years and older.
* Retired motor sport pilot (Formula 1 or rally).
* Expressing a cognitive, memory, somatic, emotional complaint, sleep disorders or a concern following the practice of Motorsport, that motivate carrying out of a memory assessment or a concussion assessment in routine care.
* Who are willing to participate in the study and give their written informed consent.
* Covered by a health insurance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retired motorsport pilots coming to the CHPG for a memory assessment or concussion assessment, meeting the study's inclusion criteria, and volunteering to participate.
  All assessments and examinations are carried out in routine care, so study essential data will be collected from the patient's medical file (source file): Demographic data, Medical history, Sport practice History of sports, Results of neurological and neuropsychological assessments, Eye-tracking results, MRI results, PET-FDG results.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Patients description | Baseline
  Describe the profile of included patients
Medical history of concussion | Baseline
  Describe the Medical history of concussion of included patients
Presence of Post Concussive Symptoms | Baseline
  Assessed by the Symptoms Scale of the Sport Concussion Assessment Tool (SCAT), composed of 22 post concussive symptom items graded on a scale from 0 (no symptoms) to 6 (severe symptoms), summed to form a symptom severity score (range 0-132).
Neurological evaluation | Baseline
  Assessed by the Neurological exam part of the Sport Concussion Assessment Tool (SCAT), composed of 5 questions.
Postural stability | Baseline
  Assessed by Balance Error Scoring System (BESS). Score of 0-60 (lower scores indicate better balance and less errors)
MRI scan | Baseline
  MRI data are described according to their nature (lesion / atrophy / sequel / signal anomaly), and classified as present or absent.
PET/CT scan - Visual analysis | Baseline
  Description of possible hypometabolic or hypermetabolic areas of the cerebral cortex on the PET / CT images of the subject.
PET/CT scan - Parametric analysis | Baseline
  The uptake values of [18F]-2-fluoro-2-deoxy-D-glucose (18-FDG) (average uptake and standard deviation) of several target regions of the subject's cerebral cortex will be entered in comparison with an age-matched database developed in the Scenium software from Siemens Medical Solutions USA® (software version VB30A)
PET/CT scan - other description | Baseline
  Description of any abnormalities found on non-opacified CT slices.
Global cognitive performance | Baseline
  MONTREAL COGNITIVE ASSESSMENT (MOCA) is used to evaluate Global cognitive performance. MOCA is a 30-question general cognitive function assessment. The maximum score is 30. Performance of each participant is compared to their reference sample (depending on age, sex and level study).
Episodic memory performance | Baseline
  The Grober and Buschke Free and Cued recall (16 items) or the Selective Reminding Test are used to evaluate Episodic memory. Performances of each participant are compared to their reference sample (depending on age, sex and level study).
Executive performance - Trail Making Test A&B | Baseline
  Trail Making Test (T.M.T) A&B is used to evaluate executive performance. The task requires a subject to connect a sequence of 25 consecutive targets on a sheet of paper, in the shortest time possible without lifting the pen from the paper. Time performances of each participant are compared to their reference sample.
Executive performance - Stroop test | Baseline
  Stroop test (GREFFEX) is used to evaluate executive performance and more specifically inhibition. The time to complete each condition (in seconds) is recorded, as well as the number of uncorrected and corrected errors. Stroop task performances of each participant are compared to their reference sample.
Executive performance - B.R.E.F. | Baseline
  The "Batterie rapide d'évaluation frontale" (B.R.E.F.), or Frontal Assessment Battery at Bedside (F.A.B.), is used to determine the presence or not of a cognitive and behavioral dysexecution syndrom. The maximum score is 18. Performances of each participant are compared to their reference sample.
Executive performance - The Modified Card Sorting Test of Nelson (MCST) | Baseline
  The Modified Card Sorting Test of Nelson (MCST) is used to evaluate executive function in patients with focal, traumatic and degenerative brain diseases. Performance on the MCST is scored by computing the number of categories achieved by a participant, and the number of perseverative errors. Performance of each participant are compared to their reference sample.
Verbal fluency | Baseline
  Verbal fluency test is a short test of verbal functioning. It consists of two tasks: category fluency and letter fluency. Participant is given 1 minute to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency). The participant's score in each task is the number of unique correct words. Performances of each participant are compared to their reference sample.
Visuospatial/constructional ability | Baseline
  Rey-complex copy figure test is used to evaluate visuospatial/constructional abilities. Performance of each participant is compared to their reference sample.
Social cognition and Emotional assessment | Baseline
  The Mini-sea is used to evaluate Social cognition. Evaluation criteria: Scores to Ekman Faces task (1976): total score / 35 and sub-scores / 5. Performances of each participant are compared to their reference sample.
Selective and sustained attention | Baseline
  The d2 Test of Attention is a cancellation test of attention and concentration that measures selective and sustained attention. Participant cross out any letter "d" with two marks around above it or below it in any order. The surrounding distractors are usually similar to the target stimulus, for example a "p" with two marks or a "d" with one or three marks (Ability to concentrate, Processing speed, Percentage of errors). The quotation provides values for the three main indices. Performances of each participant are compared to their reference sample.
Storage and handling of information, short term and working memory skill | Baseline
  The Digit span and spatial span tasks (Empans) assess the storage and handling of information, short term and working memory skill. Participant reads a sequence of numbers and is asked to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span). As well for spatial span task. Four scores are obtained (forward and backward verbal scores, forward and backward visuospatial scores). Performances of each participant are compared to their reference sample.
Working memory | Baseline
  Baddeley's dual task assess the ability to coordinate two tasks simultaneously divided attention ability. The score of each participant are compared to their reference sample.
A sustained attention and working memory test | Baseline
  PASAT (Paced Auditory Serial Addition Test) is a sustained attention and working memory test. The results are expressed as a score of 60 points. Performances of each participant are compared to their reference sample.
Language | Baseline
  The "Dénomination d'Objet 80" (DO 80), is an image naming task in order to assess language and visual gnosias.
Oculomotor paradigms raw performance - Horizontal saccades Latency | Baseline
  This concerns saccades Latency (in ms) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 Standard Deviation (SD) compared to their reference sample.
Oculomotor paradigms raw performance - Horizontal saccades Main velocity | Baseline
  This concerns saccades Main velocity (in °/sec) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 Standard Deviation (SD) compared to their reference sample.
Oculomotor paradigms raw performance - Horizontal saccades Gain. | Baseline
  This concerns saccades Gain (gaze accuracy) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 Standard Deviation (SD) compared to their reference sample.
Oculomotor paradigms raw performance - Vertical saccades Latency | Baseline
  This concerns saccades Latency (in ms) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Oculomotor paradigms raw performance - Vertical saccades Main Velocity | Baseline
  This concerns saccades Main velocity (in °/sec) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Oculomotor paradigms raw performance - Vertical saccades Gain | Baseline
  This concerns saccades Gain (gaze accuracy) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Inhibition capacity | Baseline
  Measure of inhibition capacity performance during an "antisaccades" paradigm. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: percentage of errors. For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Internuclear ophthalmoplegia (INO) detection | Baseline
  Highlight presence/absence of INO. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: INO is present if calculated ratio of abducting to adducting eye movement (both mean and peak velocity) is >1.
Fixations impairments detection | Baseline
  Highlight presence/absence of Fixations impairments. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: presence/absence/frequency of square wave-jerks, nystagmus, flutters.
Impairment of smooth pursuit | Baseline
  Highlight Impairment of horizontal and vertical smooth pursuit. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: presence/absence of saccade and perturbation.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PAULMIER, Principal Investigator — Department of Nuclear Medicine, Princess Grace Hospital, Monaco.
Locations (1):
- Princess Grace Hospital / Department of Nuclear Medicine / Memory Center of the Rainier III Clinical Gerontology Center, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No